CLINICAL TRIAL: NCT03400033
Title: A Phase 3 Randomized, Double-blind, Active-controlled, Parallel-group, Multi-center Study in Hemodialysis Participants With Anemia of Chronic Kidney Disease to Evaluate the Efficacy, Safety and Pharmacokinetics of Three-times Weekly Dosing of Daprodustat Compared to Recombinant Human Erythropoietin, Following a Switch From Recombinant Human Erythropoietin or Its Analogs
Brief Title: Anemia Studies in Chronic Kidney Disease (CKD): Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor (PHI) Daprodustat-Three-times Weekly Dosing in Dialysis (ASCEND-TD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 204837; 2017-004372-56 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Anaemia
Keywords: CKD, EPO, rhEPO, Hemodialysis dependent, Daprodustat
MeSH Terms: conditions — Anemia | interventions — GSK1278863

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either daprodustat or epoetin alfa in a parallel manner. .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study, in which the subject, investigator, site staff and the sponsor will remain blinded to each subjects study treatment assignment throughout the course of the study, with the exception of a limited number of unblinded site staff who are necessary to maintain the blind, as well as a limited number of sponsor staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daprodustat (Experimental): Subjects randomized to this arm will receive daprodustat tablets titrated doses from 2 to 48 milligrams orally three-times weekly along with saline by IV route for the 52 weeks treatment period.
  Interventions: Drug: Daprodustat tablets; Drug: Saline vials or bags
- Epoetin alfa (Active Comparator): Subjects randomized to this arm will receive matching placebo tablets to daprodustat orally three-times weekly and Epoetin alfa by IV route for the 52 weeks treatment period.
  Interventions: Drug: Matching placebo tablets; Drug: Epoetin alfa vials

INTERVENTIONS:
Drug: Daprodustat tablets — Round, biconvex, white, film-coated tablet in unit dose strengths 2 and 4 milligrams (7 millimeter tablets), 6, 8 and 10 milligrams (9 millimeter tablets) administered by the oral route.
  Arms: Daprodustat
Drug: Matching placebo tablets — Matching placebo to daprodustat tablets supplied as round, biconvex, white, film-coated tablet in unit dose strengths 2 and 4 milligrams (7 millimeter tablets), 6, 8 and 10 milligrams (9 millimeter tablets) administered by the oral route.
  Arms: Epoetin alfa
Drug: Epoetin alfa vials — Single-dose, preservative-free vials in unit dose strengths of 2000, 3000, 4000 and 10,000 Units/milliliter administered by the IV route.
  Arms: Epoetin alfa
Drug: Saline vials or bags — 0.9% sodium chloride saline vials or bags administered by the IV route.
  Arms: Daprodustat

SUMMARY:
This Phase 3 study in hemodialysis-dependent subjects with anemia will evaluate the efficacy and safety of daprodustat administered three-times weekly compared to epoetin alfa, the current standard of care. This study includes a 4 week Screening Period, a 52 week Treatment Period and a 4 to 6 week follow-up period. Each subject will remain in the study for up to 62 weeks. Approximately 402 subjects will be randomized to receive either daprodustat three times weekly or epoetin alfa three-times weekly or once weekly, depending on dose level.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 99 years of age inclusive, at the time of signing the informed consent.
* Use of any approved rhEPO or analog for at least 8 weeks prior to the screening visit and continuing during the screening period until randomization (Day 1).
* Hgb concentration (measured by HemoCue) within the following range: Week -4: Hgb 8 to 11.5 grams/deciliter (5 to 7.1 millimoles/liter). If Hgb is 11.6 to 11.9 grams/deciliter (7.2 to 7.4 millimoles/liter), up to two retests are allowed; the retest value must be between 8 to 11.5 grams/deciliter (5 to 7.1 millimoles/liter). Day 1: Hgb 8 to 11 grams/deciliter (5 to 6.8 millimoles/liter) and receiving at least the minimum rhEPO or analog dose 3. Hgb>11 to 11.5 grams/deciliter (6.8 to 7.1 millimoles/liter) and receiving greater than the minimum rhEPO or analog dose 3.
* On hemodialysis (including hemofiltration or hemodiafiltration) >90 days prior to screening and continuing during the screening period.
* On hemodialysis (in-center) >=3 times per week.
* Male and female subjects are eligible. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP), or A WOCBP who agrees to follow the contraceptive guidance from at least 28 days prior to first dose of study treatment and for at least 28 days after the last dose of study treatment.
* Capable of giving signed informed consent.
* In France, a subject will be eligible for inclusion in this study if he or she is either affiliated to or beneficiary of a social security category.

Exclusion Criteria:

* Planned living-related or living-unrelated kidney transplant within 52 weeks after randomization (Day 1).
* Ferritin: <=100 nanograms/milliliter (<=100 micrograms/liter), at screening.
* Transferrin saturation (TSAT): <=20 percent, at screening. If TSAT is 18 to 20 percent, then a retest using a new blood sample can be obtained within 7 days of the final laboratory report; the final retest value must be >20 percent to confirm eligibility.
* Aplasias: History of bone marrow aplasia or pure red cell aplasia.
* Conditions, other than anemia of CKD, which can affect erythropoiesis.
* Myocardial infarction (MI) or acute coronary syndrome within 8 weeks prior to screening through to randomization (Day 1).
* Stroke or transient ischemic attack within 8 weeks prior to screening through to randomization (Day 1).
* Heart failure (HF): Chronic Class IV HF, as defined by the New York Heart Association (NYHA) functional classification system.
* Current uncontrolled hypertension as determined by the investigator that would contraindicate the use of rhEPO.
* Bazett's correction of QTc interval (QTcB): at Day 1: QTcB >500 milliseconds, or QTcB >530 milliseconds in subjects with bundle branch block. There is no QTc (corrected QT) exclusion for subjects with a predominantly ventricular paced rhythm.
* Liver Disease: presence of any one of the following liver-related laboratory values or conditions, at screening, is exclusionary: ALT >2x upper limit of normal (ULN); Bilirubin >1.5x ULN; or Current unstable liver or biliary disease per investigator assessment, generally defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Evidence of actively bleeding gastric, duodenal or esophageal ulcer disease OR clinically significant gastro intestinal bleeding <= 8 weeks prior to screening through to randomization (Day 1).
* History of malignancy within 2 years prior to screening through to randomization (Day 1), currently receiving treatment for cancer, or complex kidney cyst (e.g., Bosniak Category IIF, III or IV) >3 centimeters.
* Use of a strong inhibitor of Cytochrome P4502C8 [CYP2C8] (e.g. gemfibrozil) or a strong inducer of CYP2C8 (e.g. rifampin/rifampicin).
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product (daprodustat) or epoetin alfa.
* Use of another investigational agent within 30 days or within five half-lives of the investigational agent (whichever is longer) or currently participating in a study of an investigational device prior to screening through to randomization (Day 1).
* Any prior treatment with daprodustat for treatment duration of >30 days.
* Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the subject at unacceptable risk, which may affect study compliance (e.g. intolerance to rhEPO) or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (83):
- United States (22):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Middlebury, Connecticut
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Pittsfield, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, College Point, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Norfolk, Virginia
- Argentina (4):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Pergamino, Buenos Aires
  - GSK Investigational Site, Sarandí, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
- Australia (2):
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Parkville, Victoria
- Brazil (7):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Passo Fundo, Rio Grande do Sul
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, São Paulo
- GSK Investigational Site, Oshawa, Ontario, Canada
- France (5):
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Epagny Metz-Tessy
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Strasbourg
- Italy (4):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Verona, Veneto
- Poland (5):
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Sandomierz
  - GSK Investigational Site, Tarnowskie Góry
  - GSK Investigational Site, Żyrardów
- Romania (2):
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Reşiţa
- Russia (14):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kolomna
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Krasnogorsk
  - GSK Investigational Site, Mytischi
  - GSK Investigational Site, Novorossiysk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Podolsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yaroslavl
- South Korea (5):
  - GSK Investigational Site, Anyang-Si, Gyeonggi-do
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (8):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Granollers, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Manises (Valencia)
  - GSK Investigational Site, Sanlúcar de Barrameda (Cádiz)
- United Kingdom (4):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, London
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Coyne DW, Singh AK, Lopes RD, Bailey CK, DiMino TL, Huang C, Connaire J, Rastogi A, Kim SG, Orias M, Shah S, Patel V, Cobitz AR, Wanner C. Three Times Weekly Dosing of Daprodustat versus Conventional Epoetin for Treatment of Anemia in Hemodialysis Patients: ASCEND-TD: A Phase 3 Randomized, Double-Blind, Noninferiority Trial. Clin J Am Soc Nephrol. 2022 Sep;17(9):1325-1336. doi: 10.2215/CJN.00550122. Epub 2022 Aug 2. PMID 35918106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 90 centers in 13 countries. Participants were randomized to receive either Daprodustat or Epoetin alfa.
Pre-assignment Details: A total of 595 participants were screened, of which 188 were screen failures. A total of 407 participants were enrolled in the study.
Groups:
- Daprodustat: Participants received daprodustat tablets with titrated dose levels ranging from 2, 4, 8, 12, 16, 20, 24, 32 and 48 milligrams (mg) orally three-times weekly up to 52 weeks. Study treatment was dose-titrated to achieve and maintain hemoglobin in the target range (10 to 11 grams per deciliter [g/dL]). In order to maintain the study blind, participants also received saline intravenous (IV) injection once weekly or three-times weekly depending on dose level, up to 52 weeks as an inactive treatment for the IV formulation. All participants were followed up at 4 to 6 weeks after last dose.
- Epoetin Alfa: Participants received epoetin alfa with titrated dose levels ranging from 1500 Units to 60,000 Units total weekly dose and administered as IV injection once weekly or three-times weekly depending on dose level up to 52 weeks. Study treatment was dose-titrated to achieve and maintain hemoglobin in the target range (10 to 11 g/dL). In order to maintain the study blind, participants also received placebo tablets matching to daprodustat orally three-times weekly up to 52 weeks as an inactive treatment for the tablet formulation. All participants were followed up at 4 to 6 weeks after last dose.
Period: Overall Study
Arm/Group | Daprodustat | Epoetin Alfa
Started | 270 | 137
Completed | 269 | 135
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat | Epoetin Alfa | Total
Number analyzed (Participants) | 270 | 137 | 407
Age, Customized [Count of Participants; unit: Participants]
  19-64 Years | 167 | 96 | 263
  >= 65 Years | 103 | 41 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 56 | 177
  Male | 149 | 81 | 230
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 49 | 32 | 81
  AMERICAN INDIAN OR ALASKAN NATIVE | 1 | 1 | 2
  ASIAN - CENTRAL/SOUTH ASIAN HERITAGE | 1 | 0 | 1
  ASIAN - EAST ASIAN HERITAGE | 16 | 9 | 25
  ASIAN - SOUTH EAST ASIAN HERITAGE | 3 | 0 | 3
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1 | 0 | 1
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 1 | 4 | 5
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 193 | 90 | 283
  MIXED WHITE RACE | 1 | 0 | 1
  MIXED RACE | 1 | 1 | 2
  UNKNOWN | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hemoglobin Levels Over the Evaluation Period (Week 28 to Week 52)
Description: Blood samples were collected from participants for hemoglobin measurements. Hemoglobin during the evaluation period was defined as the mean of all available post-randomization hemoglobin values (on and off-treatment) during the evaluation period (Week 28 to Week 52). For the primary analysis, the missing post-Baseline hemoglobin values were imputed using pre-specified multiple imputations. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date, including those from unscheduled visits. Change from Baseline was defined as the average of post-randomization values during the evaluation period minus Baseline value. Analysis was performed using the Analysis of Covariance (ANCOVA) model with terms for treatment, Baseline hemoglobin, and region.
Time Frame: Baseline (Pre-dose on Day 1) and evaluation period (Week 28 to Week 52)
Population: All Randomized (Intent-to-treat [ITT]) Population comprised of all randomized participants. Any participant who received a treatment randomization number was considered to have been randomized.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 270 | 137
Grams per deciliter (g/dL) | -0.04 (0.045) | 0.02 (0.066)
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95 percent (%) confidence interval (CI) for the treatment difference is greater than the pre-specified non-inferiority margin of -0.75 g/dL; Least square (LS) mean difference = -0.05, 95% CI 2-sided [-0.21 to 0.10]

2. Secondary Outcome: Mean Average Monthly On-treatment Intravenous (IV) Iron Dose Per Participant
Description: Average monthly IV iron dose (mg) per participant during Day 1 to Week 52 was determined by calculating the total IV iron dose per participant from Day 1 to Week 52 while the participant was on study treatment and dividing by (the number of days the participant was on study treatment divided by 30.4375 days). Analysis was performed using the ANCOVA model with terms for treatment, Baseline monthly IV iron dose, and region.
Time Frame: Day 1 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Milligrams
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 270 | 136
Milligrams | 98.11 (11.049) | 106.23 (15.569)
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.3354, ANCOVA; LS mean difference = -8.12, 95% CI 2-sided [-45.66 to 29.41]

3. Secondary Outcome: Change From Baseline in Hemoglobin Levels at Week 52
Description: Blood samples were collected from participants for hemoglobin measurements. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date, including those from unscheduled visits. Change from Baseline was defined as the post-randomization visit value minus Baseline value. Analysis was performed using a mixed model repeated measures (MMRM) model fitted to hemoglobin data collected after Baseline up to Week 52, excluding values collected during the stabilization period (Day 1 to Week 28). The model included factors for treatment, time, region, Baseline hemoglobin and Baseline hemoglobin by time and treatment by time interaction terms.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 252 | 128
Grams per deciliter | -0.03 (0.069) | 0.11 (0.098)
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% CI for the treatment difference is greater than the pre-specified non-inferiority margin of -0.75 g/dL; LS mean difference = -0.14, 95% CI 2-sided [-0.37 to 0.10]

4. Secondary Outcome: Percentage of Time With Hemoglobin in the Analysis Range (10 to 11.5 Grams/Deciliter) Over Evaluation Period (Week 28 to Week 52)
Description: Participants received treatment during the study to achieve or maintain hemoglobin level in the target range. Percentage of time for which hemoglobin level was maintained within the analysis range (10 to 11.5 grams/deciliter) has been presented.
Time Frame: Week 28 to Week 52
Population: All Randomized (ITT) Population. Only those participants with at least one evaluable hemoglobin value during the evaluation period were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percentage of days
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 215 | 107
Percentage of days | 70.83 [50.98 to 91.07] | 61.76 [29.69 to 85.19]
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% CI for the treatment difference was above the non-inferiority margin of - 15%; p = 0.0034, Van Elteren's test; Median Difference (Final Values) = 11.18, 95% CI 2-sided [2.83 to 19.56] — Hodges-Lehmann Estimate of Treatment Difference has been reported

5. Secondary Outcome: Number of Hemoglobin Responders in the Hemoglobin Analysis Range (10 to 11.5 Grams/Deciliter) Over Evaluation Period (Week 28 to Week 52)
Description: Mean hemoglobin during the evaluation period was defined as the mean of all evaluable hemoglobin values during the evaluation period (Week 28 to Week 52) including any evaluable unscheduled hemoglobin values that were taken during this time period. Hemoglobin responders were defined as the number of participants with a mean hemoglobin during the evaluation period that falls within the hemoglobin analysis range of 10-11.5 grams/deciliter.
Time Frame: Week 28 to Week 52
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 215 | 107
Participants | 172 | 68
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Other; p = 0.0007, Cochran-Mantel-Haenszel; Difference in response rate = 0.1645, 95% CI 2-sided [0.06 to 0.27]

6. Secondary Outcome: Percentage of Participants Permanently Stopping Study Treatment Due to Meeting Rescue Criteria
Description: Percentage of participants permanently stopping study treatment due to meeting rescue criteria has been presented.
Time Frame: Up to Week 52
Population: All Randomized (ITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 270 | 137
Percentage of participants | 2.2 | 2.2
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Other; p = 0.5308, Wald test; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.26 to 4.22] — Hazard ratio is estimated using a Cox proportional hazard regression model adjusted for treatment group and region

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Arterial Pressure (MAP) at Week 52
Description: Measurements for SBP, DBP and MAP were taken with the participant in a semi-supine or seated position in the dialysis chair after at least a 5-minute rest period. MAP is the average BP in an individual's arteries during a single cardiac cycle. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date, including those from unscheduled visits. Change from Baseline was defined as the on-treatment visit value minus Baseline value. Analysis was performed using MMRM model with treatment group, time, region, Baseline value, Baseline value*time, treatment group*time as variables.
Time Frame: Baseline (Week -4 ) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 266 | 133
Millimeter of mercury (mmHg)
  SBP | -3.18 (1.470) | 0.55 (2.252)
  DBP | -2.52 (0.764) | -0.29 (1.176)
  MAP | -2.72 (0.907) | -0.12 (1.389)
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.083, MMRM; LS mean difference = -3.73, 95% CI 2-sided [-9.03 to 1.56] — SBP
Statistical Analysis 2: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.057, MMRM; LS mean difference = -2.23, 95% CI 2-sided [-4.99 to 0.54] — DBP
Statistical Analysis 3: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.059, MMRM; LS mean difference = -2.60, 95% CI 2-sided [-5.86 to 0.67] — MAP

8. Secondary Outcome: Change From Baseline in SBP, DBP and MAP at End of Treatment
Description: Measurements for SBP, DBP and MAP were taken with the participant in a semi-supine or seated position in the dialysis chair after at least a 5-minute rest period. MAP is the average BP in an individual's arteries during a single cardiac cycle. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date, including those from unscheduled visits. Change from Baseline was defined as the last on-treatment visit value minus Baseline value. Analysis was performed using ANCOVA model with terms for treatment group, region and Baseline value. Adjusted mean and standard error have been presented.
Time Frame: Baseline (Week -4) and end of treatment (last on-treatment value until Week 52)
Population: All Randomized (ITT) Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 270 | 136
Millimeter of mercury (mmHg)
  SBP | -1.4 (1.24) | -0.9 (1.75)
  DBP | -1.8 (0.66) | -0.8 (0.93)
  MAP | -1.7 (0.78) | -0.8 (1.09)
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.407, ANCOVA; Mean Difference (Net) = -0.50, 95% CI 2-sided [-4.73 to 3.72] — SBP
Statistical Analysis 2: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.179, ANCOVA; Mean Difference (Net) = -1.05, 95% CI 2-sided [-3.29 to 1.19] — DBP
Statistical Analysis 3: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.261, ANCOVA; Mean Difference (Net) = -0.86, 95% CI 2-sided [-3.50 to 1.78] — MAP

9. Secondary Outcome: Blood Pressure (BP) Exacerbation Event Rate Per 100 Participant Years
Description: BP exacerbation event is defined (based on post-dialysis BP) as SBP >=25 mmHg increased from Baseline or SBP >=180 mmHg; or DBP >=15 mmHg increased from Baseline or DBP >=110 mmHg. The BP exacerbation events per 100 participant years was estimated using the Negative Binomial Model.
Time Frame: Up to 52 weeks
Population: All Randomized (ITT) Population. Only those participants with data available at specified time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant years
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 270 | 136
Events per 100 participant years | 250.45 [210.69 to 297.72] | 356.91 [280.95 to 453.41]
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Other; p = 0.0093, Negative binomial model; Ratio of exacerbation rate = 0.70, 95% CI 2-sided [0.52 to 0.94]

10. Secondary Outcome: Number of Participants With at Least One BP Exacerbation Event During the Study
Description: BP exacerbation (based on post-dialysis BP) is defined as: SBP >= 25 mmHg increased from Baseline or SBP >=180mmHg; or DBP >=15 mmHg increase from Baseline or DBP >=110 mmHg. Number of participants with at least 1 BP exacerbation event have been reported.
Time Frame: Up to 52 weeks
Population: All Randomized (ITT) Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 270 | 136
Participants | 151 | 91

11. Secondary Outcome: Change From Baseline at Weeks 8, 12, 28 and 52 in Patient Global Impression of Severity (PGI-S)
Description: The PGI-S is a 1-item questionnaire designed to assess participant's impression of disease severity of their anemia of Chronic kidney disease (CKD). It is measured on a 5-point disease severity scale ranging from 0 (absent) to 4 (very severe), higher score indicates more disease severity. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date, including those from unscheduled visits. Change from Baseline in on-treatment PGI-S scores was defined as the on-treatment visit value minus Baseline value. Analysis was performed using MMRM model fitted from Baseline up to Week 52 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions.
Time Frame: Baseline (Pre-dose on Day 1) and Weeks 8, 12, 28, 52
Population: All Randomized (ITT) Population. Only those participants with data available at specified time points were analyzed (represented as n=X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Epoetin Alfa
Number analyzed (Participants) | 270 | 137
Scores on a scale
  Week 8; n=248, 126: number analyzed (Participants) | 248 | 126
  Week 8; n=248, 126 | -0.10 (0.048) | 0.05 (0.068)
  Week 12; n=243, 120: number analyzed (Participants) | 243 | 120
  Week 12; n=243, 120 | -0.13 (0.050) | -0.01 (0.071)
  Week 28; n=211, 106: number analyzed (Participants) | 211 | 106
  Week 28; n=211, 106 | -0.07 (0.054) | 0.03 (0.077)
  Week 52; n=170, 85: number analyzed (Participants) | 170 | 85
  Week 52; n=170, 85 | -0.11 (0.063) | 0.04 (0.088)
Statistical Analysis 1: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.0323, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.32 to 0.01] — Week 8
Statistical Analysis 2: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.0921, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.29 to 0.06] — Week 12
Statistical Analysis 3: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.1291, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.29 to 0.08] — Week 28
Statistical Analysis 4: Comparison: Daprodustat vs Epoetin Alfa; Test type: Superiority; p = 0.0859, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.36 to 0.06] — Week 52

12. Secondary Outcome: Pre-dose Trough Concentration (Ctau) of Daprodustat (GSK1278863) and Its Metabolites GSK2391220 (M2), GSK2487818 (M4), GSK2506102 (M5), GSK2506104 (M3), GSK2531398 (M6) and GSK2531401 (M13)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of daprodustat (GSK1278863) and its metabolites: GSK2391220 (M2), GSK2487818 (M4), GSK2506102 (M5), GSK2506104 (M3), GSK2531398 (M6) and GSK2531401 (M13).
Time Frame: Pre-dose on Day 1; Pre-dose and at 0.5, 1, 2, 3 hours post-dose on any one post-Baseline visit day between Week 8 and Week 52
Population: Pharmacokinetic Population comprised of all randomized participants for whom a post-Baseline pharmacokinetic sample was obtained and analyzed. Only those participants with data available at specified time points were analyzed (represented as n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Groups:
- Daprodustat 2 mg: Participants received daprodustat tablets 2 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 4 mg: Participants received daprodustat tablets 4 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 8 mg: Participants received daprodustat tablets 8 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 12 mg: Participants received daprodustat tablets 12 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 16 mg: Participants received daprodustat tablets 16 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 20 mg: Participants received daprodustat tablets 20 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 24 mg: Participants received daprodustat tablets 24 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 32 mg: Participants received daprodustat tablets 32 mg orally three-times weekly at the time of the pharmacokinetic visit.
- Daprodustat 48 mg: Participants received daprodustat tablets 48 mg orally three-times weekly at the time of the pharmacokinetic visit.
Arm/Group | Daprodustat 2 mg | Daprodustat 4 mg | Daprodustat 8 mg | Daprodustat 12 mg | Daprodustat 16 mg | Daprodustat 20 mg | Daprodustat 24 mg | Daprodustat 32 mg | Daprodustat 48 mg
Number analyzed (Participants) | 8 | 20 | 51 | 59 | 45 | 28 | 16 | 3 | 3
Nanograms per milliliter
  Daprodustat; n=1, 2, 10, 18, 14, 9, 6, 3, 2: number analyzed (Participants) | 1 | 2 | 10 | 18 | 14 | 9 | 6 | 3 | 2
  Daprodustat; n=1, 2, 10, 18, 14, 9, 6, 3, 2 | 6.2400 (NA) — NA indicates that data was not available as geometric coefficient of variation could not be calculated for single participant. | 1.1207 (494.71) | 0.1786 (77.35) | 0.3727 (277.88) | 0.3443 (100.78) | 0.3871 (161.05) | 0.1621 (42.17) | 0.2768 (140.82) | 0.3486 (68.34)
  GSK2391220; n=4, 17,42, 57, 40, 25, 16, 3, 3: number analyzed (Participants) | 4 | 17 | 42 | 57 | 40 | 25 | 16 | 3 | 3
  GSK2391220; n=4, 17,42, 57, 40, 25, 16, 3, 3 | 0.8623 (241.17) | 0.5893 (255.59) | 0.6341 (123.92) | 1.1572 (184.51) | 1.1654 (191.57) | 1.1792 (168.59) | 1.4987 (136.35) | 1.6974 (6.82) | 1.3531 (19.28)
  GSK2487818; n=1, 4, 5, 20, 14, 7, 4, 3, 2: number analyzed (Participants) | 1 | 4 | 5 | 20 | 14 | 7 | 4 | 3 | 2
  GSK2487818; n=1, 4, 5, 20, 14, 7, 4, 3, 2 | 0.3620 (NA) — NA indicates that data was not available as geometric coefficient of variation could not be calculated for single participant. | 0.2867 (111.67) | 0.1594 (16.91) | 0.2996 (105.55) | 0.3027 (69.12) | 0.2868 (109.23) | 0.2585 (30.72) | 0.2414 (29.66) | 0.2111 (80.56)
  GSK2506102; n=4, 17, 45, 59, 43, 27, 16, 3, 3: number analyzed (Participants) | 4 | 17 | 45 | 59 | 43 | 27 | 16 | 3 | 3
  GSK2506102; n=4, 17, 45, 59, 43, 27, 16, 3, 3 | 0.9951 (122.94) | 0.8372 (121.27) | 0.9634 (95.99) | 1.5100 (105.50) | 1.5480 (122.95) | 1.6555 (133.94) | 3.2099 (67.36) | 1.6892 (30.44) | 1.8595 (48.36)
  GSK2506104; n=6, 17, 45, 59, 43, 27, 16, 3, 3: number analyzed (Participants) | 6 | 17 | 45 | 59 | 43 | 27 | 16 | 3 | 3
  GSK2506104; n=6, 17, 45, 59, 43, 27, 16, 3, 3 | 0.9750 (408.49) | 1.9588 (163.27) | 2.0381 (124.74) | 3.5141 (136.72) | 3.3872 (182.27) | 3.6000 (173.62) | 6.5730 (99.82) | 4.2068 (15.44) | 4.1894 (23.78)
  GSK2531398; n=2, 7, 22, 41, 33, 20, 15, 3, 3: number analyzed (Participants) | 2 | 7 | 22 | 41 | 33 | 20 | 15 | 3 | 3
  GSK2531398; n=2, 7, 22, 41, 33, 20, 15, 3, 3 | 1.1778 (20.55) | 0.6069 (271.48) | 0.2362 (76.76) | 0.4444 (144.99) | 0.3917 (169.77) | 0.3728 (197.51) | 0.3992 (153.15) | 0.3963 (16.52) | 0.2280 (56.68)
  GSK2531401; n=6, 17, 45, 59, 44, 27, 16, 3, 3: number analyzed (Participants) | 6 | 17 | 45 | 59 | 44 | 27 | 16 | 3 | 3
  GSK2531401; n=6, 17, 45, 59, 44, 27, 16, 3, 3 | 1.4466 (190.80) | 3.5579 (102.68) | 4.0910 (148.03) | 6.8137 (102.34) | 5.6037 (130.97) | 8.4611 (128.74) | 11.7372 (65.37) | 6.0453 (140.63) | 16.2584 (41.06)

13. Secondary Outcome: Maximum Observed Concentration (Cmax) of Daprodustat (GSK1278863) and Its Metabolites GSK2391220 (M2), GSK2487818 (M4), GSK2506102 (M5), GSK2506104 (M3), GSK2531398 (M6) and GSK2531401 (M13)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed (represented as n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Daprodustat 2 mg | Daprodustat 4 mg | Daprodustat 8 mg | Daprodustat 12 mg | Daprodustat 16 mg | Daprodustat 20 mg | Daprodustat 24 mg | Daprodustat 32 mg | Daprodustat 48 mg
Number analyzed (Participants) | 8 | 20 | 51 | 59 | 45 | 28 | 16 | 3 | 3
Nanograms per milliliter
  Daprodustat; n=8, 20, 49, 57, 45, 28, 16, 3, 3: number analyzed (Participants) | 8 | 20 | 49 | 57 | 45 | 28 | 16 | 3 | 3
  Daprodustat; n=8, 20, 49, 57, 45, 28, 16, 3, 3 | 44.5832 (227.65) | 51.9261 (227.59) | 113.4049 (179.69) | 143.8790 (233.09) | 126.6824 (288.50) | 212.5087 (152.47) | 290.3163 (87.39) | 197.7071 (36.53) | 310.1938 (190.69)
  GSK2391220; n=8, 19, 50, 59, 45, 28, 16, 3, 3: number analyzed (Participants) | 8 | 19 | 50 | 59 | 45 | 28 | 16 | 3 | 3
  GSK2391220; n=8, 19, 50, 59, 45, 28, 16, 3, 3 | 2.6298 (60.93) | 4.0224 (134.91) | 6.3826 (198.78) | 8.9535 (126.76) | 9.5131 (167.92) | 11.8995 (172.35) | 22.3378 (95.60) | 9.3582 (71.78) | 31.6698 (84.08)
  GSK2487818; n=7, 18, 47, 56, 45, 28, 16, 3, 3: number analyzed (Participants) | 7 | 18 | 47 | 56 | 45 | 28 | 16 | 3 | 3
  GSK2487818; n=7, 18, 47, 56, 45, 28, 16, 3, 3 | 2.0320 (73.45) | 3.2703 (143.75) | 6.3474 (175.79) | 8.0134 (146.43) | 6.4276 (278.04) | 9.6617 (207.18) | 19.9693 (94.09) | 8.4327 (64.98) | 29.3042 (72.06)
  GSK2506102; n=8, 19, 51, 59, 45, 28, 16, 3, 3: number analyzed (Participants) | 8 | 19 | 51 | 59 | 45 | 28 | 16 | 3 | 3
  GSK2506102; n=8, 19, 51, 59, 45, 28, 16, 3, 3 | 0.8328 (101.92) | 1.4018 (84.93) | 2.0385 (85.59) | 2.8357 (68.15) | 3.2007 (89.86) | 3.5712 (96.48) | 6.4555 (59.57) | 2.4981 (71.38) | 7.1245 (87.62)
  GSK2506104; n=8, 19, 51, 59, 45, 28, 16, 3, 3: number analyzed (Participants) | 8 | 19 | 51 | 59 | 45 | 28 | 16 | 3 | 3
  GSK2506104; n=8, 19, 51, 59, 45, 28, 16, 3, 3 | 3.2020 (81.23) | 5.2039 (98.70) | 7.5220 (131.81) | 10.8186 (84.31) | 11.5783 (130.74) | 13.8509 (125.27) | 24.4926 (84.96) | 9.5457 (73.58) | 30.4034 (79.13)
  GSK2531398; n=8, 17, 46, 59, 45, 27, 16, 3, 3: number analyzed (Participants) | 8 | 17 | 46 | 59 | 45 | 27 | 16 | 3 | 3
  GSK2531398; n=8, 17, 46, 59, 45, 27, 16, 3, 3 | 1.2731 (57.92) | 2.3676 (84.23) | 3.7348 (131.10) | 3.8017 (177.36) | 4.0850 (209.29) | 6.1029 (137.40) | 10.7532 (98.46) | 4.6296 (72.00) | 14.7844 (81.18)
  GSK2531401; n=7, 19, 51, 59, 45, 28, 16, 3, 3: number analyzed (Participants) | 7 | 19 | 51 | 59 | 45 | 28 | 16 | 3 | 3
  GSK2531401; n=7, 19, 51, 59, 45, 28, 16, 3, 3 | 2.0473 (100.05) | 4.0012 (88.64) | 5.4631 (120.63) | 8.8488 (80.17) | 8.4814 (93.83) | 10.7368 (90.83) | 14.7926 (59.24) | 7.1458 (174.98) | 20.1044 (67.56)

ADVERSE EVENTS:
Time Frame: Treatment emergent serious adverse events (SAEs) and non-serious adverse events (non-serious AEs) were collected up to 52 weeks.
Description: Safety Population was used to assess SAEs and non-serious AEs, which comprised of all randomized participants who have taken at least 1 dose of study treatment. One participant from Randomized (ITT) Population (N=407) did not receive study treatment, hence was not included in Safety Population (N=406).
Arm/Group | Daprodustat | Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 18/270 | 10/136
Serious Adverse Events (participants affected / at risk) | 80/270 | 47/136
Other Adverse Events (participants affected / at risk) | 74/270 | 42/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=270) | Epoetin Alfa (N=136)
Pneumonia (Infections and infestations) | 9 (9) | 5 (5)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Acinetobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Prostatitis Escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 7 (9) | 3 (4)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Extremity necrosis (Vascular disorders) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Brachiocephalic vein stenosis (Vascular disorders) | 1 (1) | 0 (0)
Dialysis induced hypertension (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (6) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Smooth muscle cell neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=270) | Epoetin Alfa (N=136)
Diarrhoea (Gastrointestinal disorders) | 23 (36) | 14 (19)
Vomiting (Gastrointestinal disorders) | 15 (16) | 13 (15)
Nausea (Gastrointestinal disorders) | 6 (8) | 11 (21)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 9 (9)
Hypertension (Vascular disorders) | 22 (35) | 14 (19)
Hypotension (Vascular disorders) | 12 (16) | 9 (13)
Pyrexia (General disorders) | 7 (9) | 8 (9)
Headache (Nervous system disorders) | 11 (13) | 13 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT03400033/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03400033/SAP_001.pdf